CLINICAL TRIAL: NCT06973278
Title: A Prospective Study on Clinical Effectiveness After SMILE Versus SMILE Xtra in Myopia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2024-267R
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMILE Group (Active Comparator)
  Interventions: Procedure: SMILE
- SMILE Xtra (Experimental)
  Interventions: Procedure: SMILE Xtra

INTERVENTIONS:
Procedure: SMILE — Small Incision Lenticule Extraction
  Arms: SMILE Group
Procedure: SMILE Xtra — Small Incision Lenticule Extraction combined with Corneal Cross-linking (SMILE Xtra)
  Arms: SMILE Xtra

SUMMARY:
To evaluate the clinical efficacy and refractive stability of SMILE Xtra compared to SMILE in patients with myopia

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 50 years.
2. High myopia with a manifest refraction spherical equivalent (MRSE) - 6.00D～-10.00D and refractive changes within ± 0.50D in the past two years;
3. Best corrected distance visual acuity (CDVA) ≥ 20/25.
4. Preoperative refractive status is stable (myopia progression not exceeding 0.50D per year for at least 2 years).
5. Predicted residual stromal thickness (RST) ≥ 250μm after lenticule removal. 6.Soft contact lenses discontinued for at least 1 week, rigid contact lenses for at least 3 weeks, and orthokeratology lenses for at least 3 months.

Exclusion Criteria:

1. The presence of other eye diseases: keratoconus or suspected keratoconus, active keratoconjunctivitis, severe dry eye, glaucoma, retinal diseases such as retinal tears or macular degeneration, etc.,
2. The presence of significant corneal scarring or cataracts affects observation.
3. Systemic diseases such as active systemic inflammation, connective tissue diseases, other conditions that prevent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
visual acuity | 1 week, 1 month, 6 months, 12 months，24 months and 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Shanghai, Shanghai Municipality, China